CLINICAL TRIAL: NCT07279402
Title: TRIMPACT: A Prospective Real-World Study of Atezolizumab Monotherapy as First-Line (Stage IV) Treatment in Patients With Non-Small Cell Lung Cancer With PD-L1 Tumor Cell Expression ≥50% and No Targetable Mutations
Brief Title: TRIMPACT: Real-World First-Line Atezolizumab Use in Stage IV NSCLC With PD-L1 ≥50%
Status: Recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Derya Kivrak salim, Associate Professor, Antalya Training and Research Hospital
Other Study IDs: MON1068.1.82
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: NSCLC Stage IV; PD-L1 Gene Mutation; Atezolizumab; Real World Study
Keywords: NSCLC, PD-L1, Atezolizumab, Real World
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atezolizumab Real-World Cohort: This observational cohort consists of patients with stage IV non-small cell lung cancer (NSCLC) who receive first-line atezolizumab in routine clinical practice. Participants are included based on real-world treatment decisions made by their physicians, and no study-mandated interventions or procedures are required. The cohort reflects patients treated according to local standards of care, allowing evaluation of real-life treatment patterns, clinical outcomes, and safety in this population.

SUMMARY:
This prospective, multicenter, real-world observational study aims to evaluate the clinical outcomes of first-line atezolizumab monotherapy in patients with stage IV non-small cell lung cancer (NSCLC) with PD-L1 tumor cell expression ≥50% and no targetable mutations. The study aim to determine how atezolizumab performs in routine clinical practice with respect to survival, treatment response, and safety outcomes in this patient population in Türkiye.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, observational study designed to generate real-world evidence on the routine first-line use of atezolizumab in patients with advanced non-small cell lung cancer (NSCLC) who exhibit high PD-L1 expression and have no targetable mutations. The study does not impose any protocol-mandated procedures or intervention requirements, and all assessments, treatments, and follow-up visits are carried out according to local standards of care at each participating center.

Data will be collected prospectively from routine medical records and will include information typically obtained during standard clinical management, such as imaging assessments, laboratory results, performance status evaluations, treatment exposure, and safety monitoring. Clinical outcomes will be analyzed to describe real-world treatment patterns, variations in clinical practice, and survival and safety trends in a national cohort. Approximately 150 patients are expected to be enrolled to ensure adequate precision in estimating long-term outcomes within this population.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Diagnosis of stage IV non-small cell lung cancer.
* Male or female patients aged 18 years or older.
* Patients who have been prescribed atezolizumab in accordance with routine clinical practice and the locally approved indication in Türkiye.
* Patients who have received up to 3 cycles of atezolizumab at the screening visit.

Exclusion Criteria:

* Patients who are not receiving atezolizumab for the treatment of lung cancer according to standard of care and the approved indication.
* Known or suspected hypersensitivity to atezolizumab.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with stage IV non-small cell lung cancer receiving first-line atezolizumab as part of routine clinical practice at participating oncology centers in Türkiye. The study population reflects real-world patients treated according to local standards of care.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  Overall survival (OS) is defined as the time from the initiation of atezolizumab treatment to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  Progression-free survival (PFS) is defined as the time from the initiation of atezolizumab treatment to the first date of objectively documented disease progression (PD) or death from any cause, whichever occurs first. Progression will be assessed by the treating physician according to local standard clinical practice or RECIST criteria when available.
Objective Response Rate (ORR) | Up to 24 months
  Objective response rate (ORR) is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) during atezolizumab treatment.
Disease Control Rate (DCR) | Up to 24 months
  Disease control rate (DCR) is defined as the proportion of patients whose best overall response is complete response (CR), partial response (PR), or stable disease (SD) during atezolizumab treatment.
Duration of Response (DoR) | Up to 24 months
  Duration of response (DoR) is defined as the time from the date of first documented complete response (CR) or partial response (PR) to the first date of objectively documented disease progression or death from any cause, whichever occurs first.
One-year Overall Survival (1-year OS) | 12 months
  One-year overall survival is defined as the incidence of death from any cause within 12 months following the initiation of atezolizumab treatment.
Incidence of Hyperprogression | Up to 24 months
  The incidence of hyperprogression is defined as the proportion of patients who exhibit rapid tumor progression after initiation of atezolizumab, according to the criteria specified in the study protocol.
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to 24 months
  The incidence, nature, and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0). Safety evaluations include monitoring and recording of AEs and SAEs, laboratory results, vital signs, and other clinically relevant assessments performed as part of routine clinical practice.

CONTACTS AND LOCATIONS:
Locations (19):
- Turkey (Türkiye) (19):
  - Afyonkarahisar Health Sciences University Hospital, Afyonkarahisar
  - Ankara Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Adnan Menderes University Faculty of Medicine Hospital, Aydin
  - Dicle University Hospital, Diyarbakır
  - Trakya University Faculty of Medicine Hospital, Edirne
  - Bahçelievler Memorial Hospital, Istanbul
  - İstanbul Medipol Mega Hospital, Istanbul
  - Ümraniye Training and Research Hospital, Istanbul
  - Marmara Üniversitesi Pendik Eğitim ve Araştırma Hastanesi, Istanbul
  - Dokuz Eylul University Faculty of Medicine Hospital, Izmir
  - Necmettin Erbakan University Meram Faculty of Medicine Hospital, Konya
  - Mersin University Faculty of Medicine Hospital, Mersin
  - Ordu State Hospital, Ordu
  - Sakarya University Faculty of Medicine Hospital, Sakarya
  - Medical Park Samsun Hospital, Samsun
  - Karadeniz Technical University Farabi Hospital, Trabzon

IPD SHARING:
Plan to Share IPD: No